CLINICAL TRIAL: NCT04820400
Title: BURN 360: Reducing Pain and Anxiety During Dressing Changes After Burn Surgery Using Virtual Reality
Brief Title: Reducing Pain and Anxiety During Dressing Changes After Burn Surgery Using Virtual Reality
Acronym: BURN-360
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BURN-360
Record Dates: First submitted 2020-10-16; First posted 2021-03-29 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative; Trauma; Burns
Keywords: Virtual Reality; Prospective Randomized Controlled Trial; Decreased drug use; Pain management
MeSH Terms: conditions — Pain, Postoperative; Wounds and Injuries; Burns; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-360 group (VR-group) (Experimental): Patients will watch a VR-360 distraction video during dressing change. The patient will be asked or helped to wear the HMD write in full at the onset of a procedure and watch the VR-360 video during the dressing change procedure. When experiencing pain, the patient may indicate the need for further analgesic medication during the procedure, the patient will be asked to push a button in their hand that will trigger a light-based signal for the nurse to provide further analgesic medication. Should their hands both be involved in the burn injury, the patient will indicate the same verbally.
  Interventions: Other: Immersive VR Video
- Control Group (standard treatment) (No Intervention): The patients will receive standard treatment and will be instructed to use the same button to indicate their pain.

INTERVENTIONS:
Other: Immersive VR Video — The VR-360 video will be custom-made for the burn patient population. Through a review of current evidence for video scenarios/patients surveys, the study team will define and implement the key components appropriate for acute procedural pain such as type, duration and severity in this patient population. Next, patients will be asked about preferred pain relief elements (e.g. individual colours, geographical locations, sounds, etc.) that would help to design a video scenario. Finally, using a Likert pain scale, patients will be asked to rate each individual descriptor that exacerbates or alleviates pain. For instance, the colour red may be associated with 'flames', 'heat' and 'burns', and thus elevated pain, the colour blue may have the opposite effect, representing 'cooling' or 'cold'.
  Combined, this information will be used to create a VR-360 video geared towards alleviating acute procedural pain in patients with burn injuries undergoing dressing changes after skin graft.
  Arms: VR-360 group (VR-group)

SUMMARY:
Burn injury and its treatment is an intensely painful experience. Most severely injured patients require numerous dressing changes and skin grafting procedures (removing skin from healthy part of the body and moving it to damaged area of the body). This procedure cause extensive pain and anxiety and many patients can become dependent on pain killers during their hospital stay and throughout rehabilitation. This can delay reintegration into society and increase the chance of opioid dependence. An effective pain management plan plays a large role in patient recovery.

In addition to the physical pain experienced by these patients, burn injury is an intensely stressful and emotional life experience. This study will use a non-drug approach to reduce pain and extensive use of pain killers (opioids) during dressing changes. In particular, the study will use an immersive (allows to experience computer-generated environment as a real world) Virtual reality (VR) distraction tool during dressing change after skin graft surgery. Individuals who will decide to participate in this study will be asked to wear headgear to view immersive 360 videos specially designed by the study team. Before and after this exposure participants will be asked to complete a measurement of their anxiety level (VAS) and rate their pain.

This study will help to determine if using VR as a distraction tool during painful dressing changes will reduce pain and anxiety, and therefore opioid medications requirements, and will rely on participants experience and adapt VR videos according to participants' response.

DETAILED DESCRIPTION:
The Ross Tilley Burn Centre (RTBC) is the largest burn care centre in Canada, admitting ~300 patients/year. Most of these severely injured patients require numerous dressing changes and skin grafting procedures which cause extensive pain and anxiety in patients already facing potential losses in terms of function and independence. Poorly managed pain can reduce patient engagement and participation in effective rehabilitation, result in chronic opioid dependence, and worsen post-traumatic stress disorder.

While burn health practitioners specialize in the use of multi-modal pharmacological approach in an attempt to reduce patients' reliance on opioid, there is an increasing recognition of the importance of non-pharmacological strategies to reduce painful procedures in hospital. A number of studies have demonstrated reductions in pain, anxiety and analgesic medications with the use of Virtual Reality (VR) during procedures in hospital. VR can be applied in a variety of ways, with considerable variations in terms of cost, efficacy, and applicability. The burn injury VR literature includes predominantly small cases/series and is lacking on using VR-360 videos as a distraction technique in burn patients. Thus, VR remains under-utilized in most burn centres locally and internationally. To address this lack of knowledge, this study proposes to use VR-360 video as a distraction tool in patients during dressing changes after skin graft surgery.

This study aims to improve burn pain management by reducing opioid requirements, pain and anxiety during painful dressing changes, while also improving patient safety and satisfaction.

The study hypothesis is that immersive virtual reality use in the burn centre will reduce the cumulative dosage of analgesia used during the first two dressing changes after skin graft surgery when compared with patients not utilizing the technology.

The primary objective of this study is to evaluate the effect of VR-360 distraction video on opioid analgesic consumption during burn dressing changes.

The secondary objectives are to investigate the effect of VR-360 on pain, requirement for conscious sedation, additive effect of multiple VR exposures, anxiety, dressing change efficiency, patient reported outcome and satisfaction. Finally, patient and staff surveys will be undertaken which will allow iterative adaptation of 3600 immersive videos to the patients' preferences optimal distraction from the painful stimuli during dressing change.

The majority of patients suffering from burn injuries are committed to undergoing long, complex treatment plans that have significant physical and emotional impact. Pain is a challenge within this population and many patients require high doses of opioids. Indeed, a sizable proportion of burn patients may still require opioids as long as three months after discharge, delaying their reintegration into society and increasing the chance of opioid dependence. VR is a strategy that helps patients alter pain behavior. This study will be the first randomized trial to apply practitioner-designed VR-videos with patient input for greatest impact. It will compare opioid use, pain scores and patient satisfaction scores between this new, state of the art intervention, and current standard practice. By demonstrating VR's 'non-pharmacologic' effectiveness to alter pain perception the study team will develop a cost-effective, accessible tool that can align with practice at Sunnybrook. Furthermore, this team-based quality improvement initiative involving nurses, social workers, physio/occupational therapy and physicians aims to introduce VR as an evidence-based innovative non-pharmacological strategy to reduce opioid requirements and optimize the use of resources, workflow, and improve staff experience in burn centres across Canada and internationally

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients anticipated to receive only one skin autograft surgery for acute burn injury at RTBC (patients may have received an allograft skin procedure prior to the autograft)
* Patients who will require inpatient stay for at least two consecutive daily dressing changes
* Patients alert and oriented, and able to watch immersive video and respond to questions

Exclusion Criteria:

* Patients on mechanical ventilation
* Patients receiving intravenous sedation
* Patients with significant face, neck or scalp burn wounds
* Patients with confirmed resistant bacteria (MRSA, CPE, VRE)
* Patients with history of significant motion sickness (i.e. occur during exposure to physical, visual and virtual motion, cybersickness, etc.) verbally declared by patient
* Patients unable to communicate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid analgesia consumption | Peri-procedural (starting 4 hours before and ending 4 hours after the dressing change)
  Cumulative opioid dose (i.e. fentanyl, hydromorphone, etc.) during the first 2 dressing change sessions in intravenous morphine equivalents (IME).
Change in opioid consumption between the first two dressing changes | Peri-procedural (starting 4 hours before and ending 4 hours after the dressing change)
  Opioid consumption over the first 2 dressing changes will be assessed between the two groups and differences will be compared between two consequent dressing change events (Dressing Change Day 1 and Dressing Change Day 2). We will also compare the cumulative doses for both dressing events.

SECONDARY OUTCOMES:
Pain assessment | Immediately before, during and after each dressing change
  Study participants will rate their pain using the Numeric Rating Scale for Pain (NRS) on a scale of 0-10 (0 for no pain; 10 for unbearable pain)
Additive effect of VR exposure on pain | 2 dressing changes: Day 1 and Day 2
  The dose difference in opioid will be calculated and compared between two consequent dressing change events.
Anxiety assessment | immediately before dressing change, during and after each dressing change (30 minutes after procedure complete)
  Participants will rate their anxiety using the Visual Analogue Scale for anxiety (VASa), a 0-10 scale where 0 is "Not at all anxious" and 10 is "Extremely anxious".
Number of participants requiring conscious sedation | assessed during the dressing procedure
  The requirement for additional intravenous sedatives: ketamine (25mg IV q 5mins with no max and/or midazolam 1mg q15min (MD clinical discretion) or fentanyl (25-50 mcg IV q5 min, maximum total dose of 250mcg)
Dressing change efficiency | immediately after dressing change procedure on the day of procedure
  The dressing nurse will complete a standardized workflow questionnaire using a 0-10 Likert scale (0 as not efficient and 10 as very efficient).
Patient satisfaction: survey | assessed after 2nd dressing change on the day of procedure
  Will be assessed with a survey asking patients subjective thoughts on the procedure experience.
Opioid use at 3 months | Assessed 3 months after the procedure
  This will be a binary outcome. Whether the patient is on prescription opioid analgesics or not at the 3-month follow-up visit.
Post-Traumatic Stress Disorder Assessment | Assessed 1) at baseline 2) after 2nd dressing procedure, 3) at discharge, 4) at 3 month follow up visit
  All participants will be asked to complete the PTSD checklist for DSM-5 (PCL-5), which asks 20 questions related to symptoms of PTSD, each of which is ranked on a 0-4 scale, where 0 is "Not at all" and 4 is "extremely".

CONTACTS AND LOCATIONS:
Overall Officials: Alan D Rogers, MD, Principal Investigator — SHSC
Locations (1):
- Sunnybrook Research Institute, Toronto, Canada